CLINICAL TRIAL: NCT04514783
Title: Healthy Tissue Preservation During Wound Debridement by Using Debritom+ Micro Water Jet Technology - a Pilot Study
Brief Title: Healthy Tissue Preservation During Wound Debridement by Using Debritom+ Micro Water Jet Technology
Acronym: Debritom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Debridment
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Wound Heal; Chronic Wound
Keywords: debridement; wound care; wound bed preparation
MeSH Terms: interventions — Debridement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 2 (Other): Use of scalpel and a spoon-shaped metal instrument (curette).
  Interventions: Other: Debridement with
- Group 1 (Experimental): Use of Debritom+ micro water jet technology
  Interventions: Device: Debridement with Debritom+ micro water jet device

INTERVENTIONS:
Device: Debridement with Debritom+ micro water jet device — Visits to the outpatient wound-care center as directed by a physician. Wound care performed by the study nurse according to the study-protocol. Each necessary wound debridement will be the same and will be as follows:
  * Removal of old dressing
  * Woundworks® 3D imaging
  * Applying analgesic if necessary
  * Applying a soaked gaze with Sodium chloride (NaCl) 0.9% solution on the wound (5 minutes)
  * Debridement using Debritom+ micro water jet technology
  * Wound cleansing with NaCl 0.9% solution
  * Woundworks® 3D imaging
  * Application of new dressing (according to the wound healing phases, medical prescription)
  In the case debridement is no more required, wound dressing change will be performed as follows:
  * Removal of old dressing
  * Woundworks® 3D imaging
  * Wound cleansing with NaCl 0.9% solution
  * Application of new dressing (according to the wound healing phases, medical prescription)
  Arms: Group 1
Other: Debridement with — Visits to the outpatient wound-care center as directed by a physician. Wound care performed by the respective study nurse according to the study-protocol. Each necessary wound debridement will be the same and will be as follows:
  * Removal of old dressing
  * Woundworks® 3D imaging
  * Applying analgesic if necessary
  * Applying a soaked gaze with NaCl 0.9% solution on the wound (5 minutes)
  * Debridement using scalpel and curette
  * Wound cleansing with NaCl 0.9% solution
  * Woundworks® 3D imaging
  * Application of new dressing (according to the wound healing phases, medical prescription)
  In the case debridement is no more required, wound dressing change will be performed as follows:
  * Removal of old dressing
  * Woundworks® 3D imaging
  * Wound cleansing with NaCl 0.9% solution
  * Application of new dressing (according to the wound healing phases, medical prescription)
  Arms: Group 2

SUMMARY:
Chronic wounds are common and carry out an important and often neglected burden not only to the individual, the family but also to the society as a whole. The therapeutic approach to the management of chronic wounds include wound bed preparation or wound dressing management. Wound bed preparation is a concept emphasizing a holistic and systematic approach to evaluate and remove barriers to the healing process to allow the wound healing process to progress normally. Debridement is an integrated part of wound bed preparation, achieving certain goals and, thus, creating a healthy wound bed, margins and peri-wound skin with the objective to promote and accelerate healing. Debridement is defined as the removal of foreign material and necrotic tissue from a wound and it can also help to stimulate wound healing. However, not all methods of debridement are the same. Each method has advantages and disadvantages that must be clearly understood. In the present clinical practice, there are several methods of wound debridement: autolytic, enzymatic, mechanical, surgical (sharp) and biologic. The most common method is the mechanical debridement. Currently a micro-water jet technique was introduced into clinical practice. The micro-water jet technique Debritom+ is an effective alternative to traditional instrument interventions performed with the scalpel and/or curette. A sterile liquid is expelled from a nozzle at a selected intensity and accurately sprayed onto the wound surface. The desired effect is the generation of targeted micro-bleedings to stimulate regeneration and healing processes while preserving the underlying healthy tissue.

Today, there is no clinical evidence quantitatively comparing one debridement method over the other. Therefore the invesitgators propose a pilot study to measure the extent of tissue loss after debridement using Debritom+ micro-water jet technology versus traditional instrument debridement procedure using scalpel and curette.

DETAILED DESCRIPTION:
Chronic wounds (CWs) are common and carry out an important and often neglected burden not only to the individual, the family but also to the society as a whole. A wound becomes chronic when they fail to progress through a timely sequence of repair resulting in anatomic and functional integrity within a period of approximatively three months. CWs affect a large segment of the world population (3) with a prevalence of mixed aetiologies of 2.21 per 1000. The annual costs of care of patients with CWs is estimated to be £6 billion for 2.2 million in the United Kingdom (UK).

In CWs a massive production of matrix molecules resulting from underlying cellular dysfunction and dysregulation can be found. Fibrinogen and fibrin are also common in chronic wounds and it is thought that these and other macromolecules scavenge growth factors and other molecules involved in promoting wound repair. Chronic wound fluid is also biochemically distinct from acute wound fluid; it slows down, and can block the proliferation of cells, which are essential for the wound healing process. The therapeutic approach to enhance the wound healing process include wound bed preparation or wound dressing management. Wound bed preparation as a concept allows the clinician to focus systematically on all of the critical components of a non-healing wound to identify the cause of the problem, and implement a care programme so as to achieve a stable wound that has healthy granulation tissue and a well vascularised wound bed. Debridement is an integrated part of wound bed preparation, achieving certain goals and, thus, creating a healthy wound bed, margins and peri-wound skin with the objective to promote and accelerate healing (8). Debridement is defined as the removal of foreign material and necrotic tissue from a wound and it can also help to stimulate wound healing (8). However, not all methods of debridement are the same. Each method has advantages and disadvantages that must be clearly understood.

In the present clinical practice, there are several methods of wound debridement: autolytic, enzymatic, mechanical, surgical (sharp) and biologic. The most common method is the mechanical debridement. Autolytic, chemical, and surgical methods are considered to be selective techniques, whereas mechanical methods are considered to be nonselective. Selective modalities remove mainly necrotic tissue, whereas nonselective modalities remove both necrotic and viable tissue. In practice, selective modalities can also remove or damage healthy tissue. The most selective modalities are autolytic and biologic techniques. Instrument debridement is the most used debridement method from many years. It has been shown to improve wound healing and its main advantages are the low cost of treatment and the speed of dead tissue removal. This method is done with the intention of removing small amounts of visible devitalized tissue. However, residual nonviable tissue may remain at the microscopic level resulting in slowing healing process. On the contrary, the risk of exaggerated / mismanaged excision is not non-existent and can lead to damage to healthy tissue or even damage to deeper structures (blood vessels, nerves, tendons or even bones), resulting in delayed healing too. Instrument debridement can be painful. Patient's fear about this approach is a reality that can also be problematic. Autolytic or enzymatic debridement, which are more selective and less prone to patient's reluctance could remediate to this situation. However, time for complete dead tissue removal is considerably increased, requiring multiple applications and stringent patient compliance. While this type of debridement does not damage healthy tissue and causes little or no pain, it can cause contact sensitization. Water-jet debridement systems seems to pose a valid alternative to other methods. The approach is based on mechanical and homogenous wound cleansing and stimulation by a micro-jet of water. It uses an ultra-fine, powerful and adjustable micro-jet of water that precisely removes soft to fibrous deposits from the wound. It is usually fast. Softness of the treatment depends on the speed and intensity of the water jet according to wound condition. Adequate pain control should be performed and surface anaesthesia may be required. Water jet debridement promotes natural wound healing by inducing micro-bleeding from the wound bed and minimizes scarring. While there is ample anecdotal evidence about the efficacy of such method to preserve healthy tissue, the investigators propose here to document this ability by measuring precisely wound depth before and after debridement using Debritom+ micro water jet technology. The investigators propose to systematically assess patient's apprehension regarding this technique too.

ELIGIBILITY:
Inclusion Criteria:

* An existing chronic wound requiring debridement
* Age over 18 years
* Proficiency in the French language

Exclusion Criteria:

* Valid informed consent is not or cannot be given
* Patients with wound presenting a dry necrosis
* Arterial insufficiency stage III or IV
* Patients under double anti-aggregation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
change in wound depth | 6 weeks
  to determine the invasiveness of each debridement technique by the measures of wound dimensions (length, width, depth, area and volume) using Woundworks® device before and after debridement over a 6 weeks treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian E Probst, Prof Dr, Study Chair — HES-SO University of Applied Sciences and Arts Western Switzerland
Locations (1):
- Cité Génération Maison de santé, Onex, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
data will be anonymised